CLINICAL TRIAL: NCT06394700
Title: Written Exposure Therapy and App-Delivered Mindfulness-Based Meditation for PTSD and Subthreshold PTSD in China: A Pilot Randomized Controlled Trial
Brief Title: Written Exposure Therapy and App-Delivered Mindfulness Meditation for PTSD in China: A Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yinyin Zang, PhD, Principal Investigator, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WET-PTSD-CN-PILOT
Record Dates: First submitted 2024-04-23; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: PTSD; Insomnia, Secondary
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders | interventions — Wettability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Written Exposure Therapy (WET) (Experimental)
  Interventions: Behavioral: written exposure therapy
- Written Exposure Therapy plus mindfulness-based App (WET+MBA) (Experimental)
  Interventions: Behavioral: Written Exposure Therapy plus Mindfulness-Based App (WET + MBA)
- Minimal Contact Control (MCC) (Placebo Comparator)
  Interventions: Behavioral: Minimal Contact Control (MCC)

INTERVENTIONS:
Behavioral: written exposure therapy — Written Exposure Therapy (WET) is a manualized exposure-based therapy involving five sequential weekly individual sessions. Each session lasts approximately 40 minutes except the first, which is one hour. In the initial session, the therapist explains the treatment rationale and guides the participant to write about their traumatic experience uninterrupted for 30 minutes. Subsequent sessions start with a brief discussion about the previous session's writing, followed by another 30-minute writing session, concluding with a short check-in. There is no homework between sessions.
  Arms: Written Exposure Therapy (WET)
Behavioral: Written Exposure Therapy plus Mindfulness-Based App (WET + MBA) — WET + MBA combines the standard WET protocol with the addition of a mindfulness practice facilitated through a mobile app called "Now Meditation." This app is among the most downloaded mindfulness apps in China, used to help manage symptoms of insomnia commonly comorbid with PTSD. Participants are instructed to engage in daily mindfulness exercises according to the app's "7-Day Basic Meditation" program and continue practicing mindfulness throughout the duration of the therapy. This is intended to supplement the therapeutic effects of WET by providing tools to manage insomnia and potentially enhancing the therapeutic process by fostering greater mindfulness and relaxation.
  Arms: Written Exposure Therapy plus mindfulness-based App (WET+MBA)
Behavioral: Minimal Contact Control (MCC) — MCC contains weekly phone calls from a study therapist to monitor their status and provide support as needed, without introducing any specific therapeutic interventions. These calls are brief, generally lasting between 10 to 15 minutes, and are strictly for the purpose of engagement and safety monitoring rather than therapeutic intervention.
  Arms: Minimal Contact Control (MCC)

SUMMARY:
The goal of this study is to use a pilot RCT to assess the effectiveness of Written Exposure Therapy (WET) and a mindfulness-based app (MBA) for managing PTSD and comorbid insomnia in China. The main questions it aims to answer are:

1. Does WET alone reduce PTSD symptoms in Chinese patients with PTSD and subthreshold PTSD?
2. Does the addition of MBA to WET lead to greater reductions in comorbid insomnia symptoms compared to WET alone?

Researchers will compare WET alone and MCC to see if WET provides benefits in managing PTSD. Researchers will compare WET plus MBA and WET group to see if the integrated MBA treatment provides additional benefits in managing insomnia.

Participants will:

* Undergo random assignment to one of three groups: WET, WET plus MBA, or MCC.
* Receive clinical interviews for primary outcomes (PTSD symptoms) at baseline, posttreatment, and during follow-ups.
* Provide self-reported data on PTSD symptoms and insomnia severity at multiple time points.
* In the WET plus MBA group, additionally use a mindfulness-based app as part of their treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and female aged between 18-65 years old;
2. A diagnosis of PTSD or subthreshold PTSD (PTSD Symptom Scale, Interview Version for DSM-5, PSSI-5);
3. If currently taking psychotropic medication, taking a stable one for at least 4 weeks;
4. A smartphone owner and no obstacle to the Now Meditation App;
5. Scoring 12 or more on Insomnia Severity Index (ISI; the symptoms appear after the diagnosis of full/subthreshold PTSD).

Exclusion Criteria:

1. A diagnosis of bipolar disorder or psychotic disorder;
2. Current substance dependence;
3. Evidence of a moderate or severe traumatic brain injury (as determined by the obstacle to comprehending the baseline screening questionnaires);
4. Serious suicidal ideation (as determined by the Scale for Suicidal Ideation);
5. Other psychiatric disorders severe enough to warrant designation as the primary disorder;
6. Taking psychotherapy for PTSD currently.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
PTSD symptom severity | Assessed at baseline, immediately post-treatment, and at 3-month follow-up periods.
  The reduction in PTSD symptoms will be measured using the PTSD Symptom Scale, Interview Version for DSM-5 (PSSI-5). This clinician-administered interview assesses the frequency and severity of PTSD symptoms using a 5-point Likert scale ranging from 0 (not at all) to 4 (very much).

SECONDARY OUTCOMES:
Insomnia Severity | Insomnia severity is assessed at baseline, weekly during the 5-week treatment period, and at the immediate post-treatment, and 3-month follow-up assessments.
  The reduction in the severity of insomnia symptoms will be assessed using the Insomnia Severity Index (ISI). This 7-item self-report measurement evaluates the severity of insomnia symptoms, the level of satisfaction with sleep, interference with daily functioning, noticeability of impairment attributed to sleep problems, and the level of distress caused by the sleep disturbance. Each item is rated on a 5-point scale, providing a comprehensive measure of insomnia severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided